CLINICAL TRIAL: NCT05419375
Title: Master Screening Study to Determine Biomarker Status and Potential Trial Eligibility for Patients With Malignant Tumors
Brief Title: Screening Study for Participants With Malignant Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BX43361
Record Dates: First submitted 2022-06-13; First posted 2022-06-15 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-Small Cell Lung Cancer (NSCLC) (Other): Participants with NSCLC will be screened for biomarker eligibility for a linked Roche study.
  Interventions: Other: Screening platform

INTERVENTIONS:
Other: Screening platform — The screening platform will be used to determine biomarker eligibility for a linked Roche study based on tissue-based testing.

SUMMARY:
The study objective is to determine the biomarker status of a participant's tumor tissue and use that status to determine eligibility for a linked Roche clinical trial.

ELIGIBILITY:
General Inclusion Criteria:

* Confirmed availability of a representative formalin-fixed, paraffin-embedded (FFPE) tumor specimen meeting criteria defined in the protocol
* Considered by principal investigator (PI) to be a candidate for a linked clinical trial with an investigational medicinal product, and that the participant has the awareness and willingness to participate in said trial

Inclusion Criteria for Participants with Stage III NSCLC

* Locally advanced, unresectable Stage III NSCLC of either squamous or non-squamous histology based on 8th edition of the American Joint Committee on Cancer (AJCC) and Union for International Cancer Control (UICC) cancer staging system
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2

Inclusion Criteria for Participants with Stage II, IIIA, or Select IIIB (T3N2 only) NSCLC Requiring Adjuvant Treatment

* Stage II, IIIA, or select IIIB (T3N2 only) NSCLC based on the 8th edition of the AJCC and UICC cancer staging system (Amin et al. 2017)
* Considered eligible for curative intent surgery (complete resection with all surgical margins testing negative for tumor)
* Screening within Study BX43361, using a pretreatment biopsy, is encouraged to be performed as early in the participant treatment pathway as possible to ensure the participant is potentially eligible for all cohorts, and should meet guidelines as defined by the protocol
* Representative FFPE tumor specimen obtained prior to the start of any treatment
* ECOG Performance Status of 0 or 1

General Exclusion Criteria:

* History of malignancy other than NSCLC within 5 years prior to screening, except for malignancies with a negligible risk of metastasis or death
* Any condition that may affect the interpretation of study results
* Significant liver or cardiovascular disease
* Prior allogenic stem-cell or solid-organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Actual)
Dates: Start 2022-07-22 (Actual); Primary Completion 2025-09-03 (Actual); Study Completion 2025-09-03 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with evaluable biomarker results | Up to 10 years
Proportion of participants eligible for a linked Roche clinical trial | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (79):
- United States (5):
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Texas Oncology, P.A., Austin, Texas
  - Texas Oncology- Northeast Texas, Tyler, Texas
  - Oncology & Hematology Associates of Southwest Virginia, Inc, Blacksburg, Virginia
  - Northwest Cancer Specialists, Vancouver, Washington
- One Clinical Research, Nedlands, Western Australia, Australia
- Brazil (6):
  - COT - Centro Oncologico do Triangulo, Uberlândia, Minas Gerais
  - Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre X, Porto Alegre, Rio Grande do Sul
  - Clínica de Oncologia Reichow, Blumenau, Santa Catarina
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
  - Oncoclinicas Rio de Janeiro S.A., Rio de Janeiro
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada
- Chile (2):
  - Centro de Estudios Clínicos SAGA, Santiago
  - RedSalud Vitacura, Santiago
- Colombia (3):
  - Clinica De La Costa, Barranquilla
  - Hospital Universitario San Ignacio, Bogotá
  - Instituto Cancerología Medellin, Medellín
- Costa Rica (2):
  - Clinica CIMCA, San José
  - ICIMED Instituto de Investigación en Ciencias Médicas, San José
- France (2):
  - Centre Leon Berard, Lyon
  - Hia Sainte Anne, Toulon
- Germany (2):
  - Klinikum rechts der Isar der TU Muenchen, München
  - Asklepios Klinik Gauting, München-Gauting
- Queen Mary Hospital, Hong Kong, Hong Kong
- Medanta -The Medicity, Gurgaon, Haryana, India
- Rambam Medical Center, Haifa, Israel
- Azienda Ospedaliera San Camillo Forlanini, Rome, Lazio, Italy
- Japan (9):
  - Aichi Cancer Center Hospital, Aichi
  - Kobe City Medical Center General Hospital, Hyōgo
  - National Hospital Organization Himeji Medical Center, Hyōgo
  - Kagoshima University Hospital, Kagoshima
  - Kindai University Hospital, Ōsaka-sayama
  - Shizuoka Cancer Center, Shizuoka
  - Komagome Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
  - Tottori University Hospital, Tottori
- Mexico (2):
  - Clinstile S.A de C.V., Mexico City, Mexico CITY (federal District)
  - Centro de Investigación Oncologica Galerias, Aguascalientes
- Maastricht University Medical Center, Maastricht, Netherlands
- Auckland City Hospital, Cancer and Blood Research, Auckland, New Zealand
- Dolno?l?skie Centrum Chorób P?uc we Wroc?awiu, Wroc?aw, Poland
- Serbia (4):
  - University Clinical Centre of Serbia, Belgrade
  - Hospital Medical Center Bezanijska kosa, Belgrade
  - Institute for pulmonary diseases of Vojvodina, Kamenitz
  - Univ Clinical Center Kragujevac, Kragujevac
- Tan Tock Seng Hospital, Singapore, Singapore
- South Korea (6):
  - Pusan National University Yangsan Hospital, Gyeongsangnam-do
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Seoul National University Bundang Hospital, Seongnam-si
  - Kangbuk Samsung Hospital, Seoul
  - Asan Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
- Hospital Regional Universitario Carlos Haya, Málaga, Spain
- Taiwan (7):
  - National Cheng Kung Univ Hosp, Tainan
  - National Taiwan Uni Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Taipei Municipal Wan Fang Hospital, Taipei
  - Chang Gung Memorial Hospital - Linkou, Taoyuan District
  - Taichung Veterans General Hospital, Xitun Dist.
- Thailand (7):
  - National Cancer Institute, Bangkok
  - Rajavithi Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Oncology Unit, Faculty of Medicine, Vajira Hospital, Dusit
  - Srinagarind Hospital, Khon Kaen
  - Central Chest Institute of Thailand, Nonthaburi
  - Songklanagarind Hospital, Songkhla
- Turkey (Türkiye) (10):
  - Ataturk Sanatoryum Egitim Ve Arastirma Hastanesi, Ankara
  - Gazi Uni Medical Faculty Hospital, Ankara
  - Liv Hospital Ankara, Ankara
  - Bakirkoy Dr. Sadi Konuk Egitim ve Arastirma Hastanesi, Tibbi Onkoloji, Bakirkoy / Istanbul
  - Dicle University Faculty of Medicine, Diyarbakır
  - Ataturk University Medical Faculty Yakutiye Research Hospital Medical Oncology Department, Erzurum
  - Medipol University Medical Faculty, Istanbul
  - Marmara Uni Faculty of Medicine, Istanbul
  - Medikal Park Samsun, Samsun
  - Medical Park Seyhan Hospital, Seyhan
- Barts & London School of Med, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing